CLINICAL TRIAL: NCT01979874
Title: The Effects of Omega-3 Fatty Acids Supplementation on Endothelial Function and Inflammation II
Brief Title: The Effects of Omega-3 Fatty Acids on Peripheral Arterial Disease II
Acronym: OMEGA-PAD II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-11778
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pro-Omega (Experimental): High-dose, short-duration dietary omega-3 fatty acids supplementation; 325mg of EPA and 225mg of DHA per capsule. 4.4gm/day x 3 months (Nordic Naturals, Watsonville, CA, USA)
  Interventions: Dietary Supplement: Pro-Omega
- Placebo (Placebo Comparator): Pro-Omega Placebo soybean capsules (Nordic Naturals, Watsonville, CA, USA); 4.4gm/day x 3 months
  Interventions: Other: ProOmega Placebo

INTERVENTIONS:
Dietary Supplement: Pro-Omega — Pro-Omega (Nordic Naturals, Watsonville, CA, USA). Each ProOmega capsule contains 325mg of EPA and 225mg of DHA. 4.4gm/day x 3 months
  Arms: Pro-Omega
Other: ProOmega Placebo — Placebo Comparator: soybean (Nordic Naturals, Watsonville, CA, USA); 4.4gm/day x 3 months
  Arms: Placebo

SUMMARY:
Investigators hypothesize that high-dose n-3 polyunsaturated fatty acids (PUFA) oral supplementation will improve systemic inflammation, vascular function, and symptomatic status of patients with PAD. Investigators will explore novel mechanistic pathways by which n-3 PUFA affect PAD, evaluating the role of specialized lipid mediators involved in the resolution of inflammation.

DETAILED DESCRIPTION:
The OMEGA-PAD II trial will be a 1:1 randomized, double-blinded trial comparing oral supplementation of n-3 PUFA (4.4g/day) to placebo in claudicants (Rutherford stage 1-3) for 3 months. Eligible patients will be screened according to specified inclusion and exclusion criteria. All patients will be treated per our current practice as reflected in the American Heart Association Practice guidelines on PAD. Blood draws, vascular function testing and 6-minute walking tests will be performed at baseline and after 3 months. n-3 PUFA supplementation will be achieved with 4 capsules of Pro-Omega twice daily (Nordic Naturals, Watsonville, California, USA), corresponding to a total of 4.4g/day. Each ProOmega capsule contains 325mg of EPA and 225mg of DHA. The placebo group will take the same number of capsules containing inactive substance (soybean; Nordic Naturals), designed to be the same color and shape as the treatment capsules.

ELIGIBILITY:
Inclusion Criteria:

1. Intermittent claudication (Rutherford 1-3)
2. One of the following:

   1. Resting or exercise ankle-brachial index (ABI) <0.9
   2. toe pressure < 70 mm Hg
   3. documentation on imaging of greater than or equal to 50% stenosis in segments of aortoiliac arteries, femoral arteries, or tibial arteries
3. Age 50 and more

Exclusion Criteria:

1. Critical limb ischemia
2. Hypersensitivity/allergies to fish or seafood
3. Already on n-3 PUFA or equivalent
4. Significant renal, hepatic, and inflammatory disease
5. Concurrent severe infections
6. Acute illness (myocardial infarction, stroke, major surgery within 30 days)
7. Receiving immunosuppressive medications or steroids
8. Age < 50

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Systemic Inflammatory bio-markers | 3 months
  reduce circulating pro-inflammatory markers (PIMs) and increase pro-resolution mediators (PRMs) assayed using targeted metabolo-lipidomics, increase PRM production within peripheral circulating monocytes.

SECONDARY OUTCOMES:
Endothelial Function | 3 months
  Will increase brachial artery flow-mediated vasodilation (FMD)and peripheral resistance (AiX) and decrease arterial stiffness in the lower extremities (PWV).

OTHER OUTCOMES:
Walking Performance | 3 months
  Will improve walking distance during 6-minute walk test and improve parameters on the walking impairment questionnaire (WIQ).

CONTACTS AND LOCATIONS:
Overall Officials: Warren Gasper, MD, Principal Investigator — UCSF & SFVAMC
Locations (1):
- San Francisco Veterans Affairs Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] Grenon SM, Hughes-Fulford M, Rapp J, Conte MS. Polyunsaturated fatty acids and peripheral artery disease. Vasc Med. 2012 Feb;17(1):51-63. doi: 10.1177/1358863X11429175. PMID 22363018
- [Background] Grenon SM, Aguado-Zuniga J, Hatton JP, Owens CD, Conte MS, Hughes-Fulford M. Effects of fatty acids on endothelial cells: inflammation and monocyte adhesion. J Surg Res. 2012 Sep;177(1):e35-43. doi: 10.1016/j.jss.2012.04.010. Epub 2012 Apr 27. PMID 22572621
- [Background] Grenon SM, Conte MS, Nosova E, Alley H, Chong K, Harris WS, Vittinghoff E, Owens CD. Association between n-3 polyunsaturated fatty acid content of red blood cells and inflammatory biomarkers in patients with peripheral artery disease. J Vasc Surg. 2013 Nov;58(5):1283-90. doi: 10.1016/j.jvs.2013.05.024. Epub 2013 Jul 2. PMID 23830313
- [Background] Grenon SM, Owens CD, Alley H, Chong K, Yen PK, Harris W, Hughes-Fulford M, Conte MS. n-3 Polyunsaturated fatty acids supplementation in peripheral artery disease: the OMEGA-PAD trial. Vasc Med. 2013 Oct;18(5):263-74. doi: 10.1177/1358863X13503695. Epub 2013 Sep 19. PMID 24052491
- See also: UCSF & SFVAMC Divisions of Vascular and Endovascular Surgery Clinical Trials — http://vascular.surgery.ucsf.edu/research/clinical-research/clinical-trials.aspx